CLINICAL TRIAL: NCT01882842
Title: The Efficacy of Endometrial Biopsy on the Outcome of In Vitro Fertilization (IVF) /Intra-Cytoplasmic Sperm Injection (ICSI) Treatment (Endoscratch): A Feasibility Pilot Study
Brief Title: A Study to Assess if Scratching the Lining of the Womb Prior to IVF Treatment Increases the Chances of Pregnancy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University of Nottingham (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12GY005
Record Dates: First submitted 2013-06-03; First posted 2013-06-20 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Infertility
Keywords: Infertility; Endometrium; Live birth
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endometrial biopsy arm (Experimental): Participants randomised to this arm arm will undergo an endometrial biopsy procedure using Pipelle endometrial sampler (Pipelle de Cornier, Laboratoire CCD, Paris, France) or Wallace/ Wallach endometrial sampler as an alternative device on cycle day LH+7 to LH+9 of the cycle directly preceding commencement of down-regulation prior to IVF or ICSI treatment. A transvaginal ultrasound scan will be performed prior to the biopsy.
  Interventions: Procedure: Endometrial biopsy; Device: Transvaginal ultrasound
- Control group (No Intervention): Participants randomised to control group will undergo a transvaginal ultrasound scan on day LH+7 to LH+9 of the cycle directly preceding commencement of IVF/ICSI treatment.

INTERVENTIONS:
Procedure: Endometrial biopsy — Endometrial biopsy will be performed in the study group and timed according to a positive urinary LH (ovulation) kit at LH+7 to +9 days.
  Other Names: Pipelle de Cornier (CCD, Paris).
  Arms: Endometrial biopsy arm
Device: Transvaginal ultrasound — A detailed assessment of the endometrium will be performed including two- and three- dimensional ultrasound, as well as power Doppler acquisitions.
  Other Names: GE Voluson E8 (Austria)
  Arms: Endometrial biopsy arm

SUMMARY:
This study aims to see if taking a small sample from the lining of the womb (the 'scratch') before starting in vitro fertilization (IVF) treatment can influence the chance of getting pregnant and having a healthy, term baby.

This study also aims to explore why an embryo is not accepted or indeed rejected by the lining of the womb. This will be analysed by carefully looking at the sample taken from the lining of the womb under the microscope and analysing the levels of natural killer (NK) cells. These cells are thought to regulate the implantation process and to be altered in some women with infertility and miscarriage.

DETAILED DESCRIPTION:
Following consent, participants will be randomised to one of the two trial interventions (endometrial biopsy, or ultrasound scan only = no intervention) by a member of the research team. The procedures will be scheduled for luteinising hormone (LH) day +7 to +9 of the menstrual cycle directly preceding commencement of down-regulation medications. A urine pregnancy test will be performed before the studied procedure. Just prior to the biopsy and directly following it, a transvaginal ultrasound scan will be performed to assess the length of the uterine cavity and endometrial parameters, including blood flow characteristics using power Doppler imaging. Endometrial sample will be obtained using standard sampling procedure by appropriately trained clinician.

Participants randomised to treatment arm will undergo an endometrial biopsy procedure using Pipelle endometrial sampler (Pipelle de Cornier, Laboratoire CCD, Paris, France) or Wallace/ Wallach endometrial sampler as an alternative device on cycle day LH+7 to LH+9 of the cycle directly preceding commencement of down-regulation prior to IVF or ICSI treatment. The endometrial sampling will be repeated a maximum of four times (all during the same appointment on day LH+7 to LH+9 of menstrual cycle) to assure a sufficient sample is obtained. If following the first two attempts, the endometrial sample is sufficient, procedure will be deemed complete. The Pipelle sampler will be introduced up to the uterine fundus (based on clinical touch technique and ultrasound measurements), and attempts will be made to obtain samples from all four walls of the endometrial cavity.

Participants randomised to control group will also be supplied with home LH testing kits after informing the unit of the will to participate. Once the ovulation test is positive, the participant will contact the unit to arrange the ultrasound appointment on day LH+7 to LH+9 of the cycle directly preceding commencement of IVF/ICSI treatment. 48 to 72 hours later and additional appointment will be scheduled for ultrasound scan and blood tests.

Subjects will then be randomised to one of the two treatment arms based on a computer generated pseudo-random code using random permuted blocks of randomly varying size, created by the University of Nottingham Clinical Trials Unit (CTU). As a pilot feasibility study, the randomisation will not be stratified by any factors. Allocation to treatments will be in the ratio 1:1. The corresponding treatment allocation will be transmitted to the unblinded clinician, who will arrange the appropriate appointments for study procedures.

Due to the nature of the study, no blinding of participant or researchers is possible.

ELIGIBILITY:
Inclusion Criteria:

* Women with history of primary or secondary infertility undergoing fresh IVF/ ICSI treatment or frozen embryo replacement cycle
* Age <49

Exclusion Criteria:

* Non- ovulatory cycles
* Absent uterus
* Uterine instrumentation within previous 3 menstrual cycles
* Women in the oocyte donation program

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
A difference in the term (37 completed weeks of gestation), singleton live birth rate in women undergoing IVF/ICSI treatment following endometrial biopsy versus control subjects. | Approximately 9 months after completion of the last procedure of the last study participant.

SECONDARY OUTCOMES:
A difference in the live birth rate (birth of a live baby after 24th week of gestation and before 37th completed weeks) in women undergoing IVF/ICSI treatment following endometrial biopsy versus control subjects. | Approximately 9 months after completion of the last procedure of the last study participant.
A difference in the multiple pregnancy rate in women undergoing IVF/ICSI treatment following endometrial biopsy versus control subjects. | Approximately 9 months after completion of the last procedure of the last study participant.
A difference in the implantation rate in women undergoing IVF/ICSI treatment following endometrial biopsy versus control subjects. | Approximately 9 months after completion of the last procedure of the last study participant.
A difference in the biochemical pregnancy rate in women undergoing IVF/ICSI treatment following endometrial biopsy versus control subjects. | Approximately 9 months after completion of the last procedure of the last study participant.
A difference in the clinical pregnancy rate in women undergoing IVF/ICSI treatment following endometrial biopsy versus control subjects. | Approximately 9 months after completion of the last procedure of the last study participant.
A difference in the miscarriage rate (loss of pregnancy before viability) in women undergoing IVF/ICSI treatment following endometrial biopsy versus control subjects. | Approximately 9 months after completion of the last procedure of the last study participant.
A difference in the ectopic pregnancy rate in women undergoing IVF/ICSI treatment following endometrial biopsy versus control subjects. | Approximately 9 months after completion of the last procedure of the last study participant.

OTHER OUTCOMES:
Sonographic markers of endometrial receptivity | Approximately 2 years
  Detailed endometrial assessment will be performed using two-, three- dimensional ultrasound, as well as power and pulse-wave Doppler ultrasound imaging. Results of these measurements will be correlated with subsequent IVF/ICSI treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Raine-Fenning, PhD, Study Chair — University of Nottingham
Locations (1):
- Nurture Fertility, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Derived] Lensen SF, Armstrong S, Gibreel A, Nastri CO, Raine-Fenning N, Martins WP. Endometrial injury in women undergoing in vitro fertilisation (IVF). Cochrane Database Syst Rev. 2021 Jun 10;6(6):CD009517. doi: 10.1002/14651858.CD009517.pub4. PMID 34110001